CLINICAL TRIAL: NCT01786629
Title: BLI800-480: A Safety and Efficacy Evaluation of 2 Different Bowel Cleansing Preparations in Adult Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Braintree Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BLI800-480
Record Dates: First submitted 2013-02-06; First posted 2013-02-08 (Estimated); Results first posted 2014-08-06 (Estimated); Last update posted 2014-08-08 (Estimated); Status verified 2014-08

CONDITIONS: Colonoscopy; Bowel Preparation; Endoscopy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SUPREP Bowel Prep Kit (Experimental): SUPREP Bowel Prep Kit
  Interventions: Drug: SUPREP Bowel Prep Kit
- FDA approved bowel preparation (Active Comparator): FDA approved bowel preparation containing electrolytes
  Interventions: Drug: FDA approved bowel preparation containing electrolytes

INTERVENTIONS:
Drug: SUPREP Bowel Prep Kit — solution for oral administration prior to colonoscopy
  Arms: SUPREP Bowel Prep Kit
Drug: FDA approved bowel preparation containing electrolytes — solution for oral administration prior to colonoscopy
  Arms: FDA approved bowel preparation

SUMMARY:
To compare the safety, tolerance and efficacy of SUPREP Bowel Prep Kit to an FDA approved control as bowel preparations prior to colonoscopy in adult patients.

ELIGIBILITY:
Inclusion Criteria:

Male or female outpatients who are undergoing colonoscopy for a routinely accepted indication.

At least 18 years of age

If female, and of child-bearing potential, is using an acceptable form of birth control

Negative urine pregnancy test at screening, if applicable

In the Investigator's judgment, subject is mentally competent to provide informed consent to participate in the study

Exclusion Criteria:

Subjects with known or suspected ileus, severe ulcerative colitis, gastrointestinal obstruction, gastric retention, bowel perforation, toxic colitis or megacolon.

Subjects who had previous significant gastrointestinal surgeries

Subjects with uncontrolled pre-existing electrolyte abnormalities, or those with clinically significant electrolyte abnormalities based on screening laboratory results, such as hypernatremia, hyponatremia, hyperphosphatemia, hypokalemia, hypocalcemia, dehydration, or those secondary to the use of diuretics or angiotensin converting enzyme (ACE) inhibitors.

Subjects with a prior history of renal, liver or cardiac insufficiency

Subjects with impaired consciousness that predisposes them to pulmonary aspiration.

Subjects undergoing colonoscopy for foreign body removal and/or decompression.

Subjects who are pregnant or lactating, or intending to become pregnant during the study.

Subjects of childbearing potential who refuse a pregnancy test.

Subjects allergic to any preparation components.

Subjects who, in the opinion of the Investigator, should not be included in the study for any reason, including inability to follow study procedures.

Subjects who have participated in an investigational surgical, drug, or device study within the past 30 days.

Subjects who withdraw consent before completion of Visit 1 procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 338 (Actual)
Dates: Start 2012-12; Primary Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John McGowan, MPH, Study Director — Braintree Laboratories, Inc.
Locations (10):
- United States (10):
  - University of South Alabama, Mobile, Alabama
  - Anaheim Clinical Trials, Anaheim, California
  - Indiana University Medical Center, Indianapolis, Indiana
  - Commonwealth Clinical Studies, Brockton, Massachusetts
  - Gastrointestinal Associates, Jackson, Mississippi
  - Long Island GI Research Group, Great Neck, New York
  - Wake Research Associates, Raleigh, North Carolina
  - Northwest Gastroenterology Clinic, Portland, Oregon
  - Franklin Gastroenterology, Franklin, Tennessee
  - Charlottesville Medical Research, Charlottesville, Virginia

REFERENCES:
- [Derived] Rex DK, DiPalma JA, McGowan J, Cleveland Mv. A comparison of oral sulfate solution with sodium picosulfate: magnesium citrate in split doses as bowel preparation for colonoscopy. Gastrointest Endosc. 2014 Dec;80(6):1113-23. doi: 10.1016/j.gie.2014.05.329. Epub 2014 Jul 12. PMID 25028274

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SUPREP Bowel Prep Kit | FDA Approved Bowel Preparation
Started | 169 | 169
Completed | 169 | 164
Not Completed | 0 | 5
Not completed — Lack of Efficacy | 0 | 4
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline Participants represents the population that was dispensed a preparation and took any portion of the preparation.
Groups:
- Total: Total of all reporting groups
Arm/Group | SUPREP Bowel Prep Kit | FDA Approved Bowel Preparation | Total
Number analyzed (Participants) | 169 | 169 | 338
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.9 (10.4) | 57.8 (9.6) | 57.8 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94 | 93 | 187
  Male | 75 | 76 | 151
Region of Enrollment [Number; unit: participants]
  United States | 169 | 169 | 338
Weight [Mean (Standard Deviation); unit: lbs] | 188 (39) | 192 (49) | 190 (45)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With a Successful Preparation (Cleaning Rated as "Good" or "Excellent")
Time Frame: Day of colonoscopy
Population: The analysis population contains subjects that consumed any portion of their bowel preparation. Subject who discontinued from the study for reasons other safety of efficacy are not included (e.g. insurance issues).
Measure: Number; unit: percentage of subjects
Arm/Group | SUPREP Bowel Prep Kit | FDA Approved Bowel Preparation
Number analyzed (Participants) | 169 | 169
percentage of subjects | 95 | 86

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events were collected for Preparation Day 1 and Day 2 (Day of Colonoscopy). Serious adverse events were collected for a period of 30 days.
Description: Adverse events for stomach cramping, stomach bloating and nausea were documented only if the symptom required an intervention or resulted in discontinuation of the bowel preparation.
Arm/Group | SUPREP Bowel Prep Kit | FDA Approved Bowel Preparation
Serious Adverse Events (participants affected / at risk) | 0/169 | 2/169
Other Adverse Events (participants affected / at risk) | 0/169 | 0/169
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SUPREP Bowel Prep Kit (N=169) | FDA Approved Bowel Preparation (N=169)
cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1)
chest pain (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 360 days from the time submitted to the sponsor for review. The sponsor cannot extend the embargo.